CLINICAL TRIAL: NCT01178450
Title: A Prospective, Randomized Trial to Compare Subtotal Parathyroidectomy Versus Cinacalcet in the Treatment of Persistent Secondary Hyperparathyroidism Post Renal Transplantation
Brief Title: Parathyroidectomy vs Cinacalcet in the Treatment of Secondary Hyperparathyroidism Post Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Josep M Cruzado (Other)
Responsible Party: Sponsor-Investigator, Josep M Cruzado, Nephrologist, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01PTHi; 2008-007017-76 (EudraCT Number)
Record Dates: First submitted 2010-04-19; First posted 2010-08-10 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Renal transplant; Hypercalcemia
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hypercalcemia | interventions — Parathyroidectomy; Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subtotal parathyroidectomy (Active Comparator): The procedure of choice is subtotal parathyroidectomy if the intraoperative biopsy confirms multiglandular disease and at least 3 glands are removed leaving a remanent of one normal gland
  Interventions: Procedure: Subtotal parathyroidectomy
- Cinacalcet (Experimental): Cinacalcet is initiated at a dose of 30 mg per day PO, adjusting the dose monthly (up to 90 mg per day PO) to achieve normocalcemia
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Procedure: Subtotal parathyroidectomy — The procedure of choice is subtotal parathyroidectomy if the intraoperative biopsy confirms multiglandular disease and at least 3 glands are removed leaving a remanent of one normal gland
  Other Names: Parathyroidectomy
  Arms: Subtotal parathyroidectomy
Drug: Cinacalcet — Cinacalcet is initiated at a dose of 30 mg per day PO, adjusting the dose monthly (up to 90 mg per day PO) to achieve normocalcemia
  Arms: Cinacalcet

SUMMARY:
The hypothesis of this study is that subtotal parathyroidectomy using minimally invasive surgery is superior to cinacalcet for the treatment of persistent secondary hyperparathyroidism (HPT) post renal transplant, with minimal morbidity and significantly reduces the cost of treatment post transplant.

DETAILED DESCRIPTION:
Persistent hyperparathyroidism (HPT) with hypercalcemia is prevalent after transplant (affects up to 25% of patients) and negatively affects graft and patient outcome. The subtotal parathyroidectomy is the standard treatment, although currently has been replaced by the calcimimetic cinacalcet. Several studies guarantee that cinacalcet is effective in controlling hypercalcemia derived of persistent HPT after renal transplantation. However, maintenance treatment is need because hypercalcemia increases quickly after treatment is stopped. This fact makes increase a lot the cost of transplantation in these patients.

The hypothesis of this study is that subtotal parathyroidectomy by minimally invasive surgery is superior to cinacalcet for treatment of persistent secondary HPT post renal transplant, with minimal morbidity and significantly reduces the cost of treatment after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Functioning renal transplant, GFR ≥ 30 ml / min
* Time post-transplant> 6 months
* PTHi>15pmol/L
* Calcium ≥2.63 mmol/L con phosphatemia ≤1.2 mmol/L
* Cervical scintigraphy
* Signed informed consent

Exclusion Criteria:

* Contraindication to surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in blood calcium levels | 12 months
  Change from baseline in blood calcium levels at 12 months.

SECONDARY OUTCOMES:
Change in parathyrin blood levels | 12 months
  Change from baseline in parathyrin blood levels at 12 months.
Patient and graft survival | 12 months
  Patient and graft survival between inclusion and month 12.
Economic evaluation of interventions measured by money spend in it. | 12 months
  Comparison of economic evaluations of both interventions between inclusion and month 12.
Estimated glomerular filtration rate. | 12 months
  Change from baseline in glomerular filtration rate at 12 months.
Change in blood calcium levels | 3 months
  Change from baseline in blood calcium levels at 3 months.
Change in blood calcium levels | 6 months
  Change from baseline in blood calcium levels at 6 months.
Change in parathyrin blood levels | 3 months
  Change from baseline parathyrin blood levels at 3 months.
Change in parathyrin blood levels | 6 months
  Change from baseline parathyrin blood levels at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Cruzado, MD, Study Chair — Nephrology Department. Hospital Universitari de Bellvitge; Pablo Moreno, MD, Study Chair — Surgery Department. Hospital Universitari de Bellvitge
Locations (2):
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelone